CLINICAL TRIAL: NCT07026968
Title: A Multicenter, Randomized, Double-blind, Parallel-controlled, Phase III Clinical Trial to Evaluate the Efficacy and Safety of the Triple Combination Therapy of Prusogliptin , Dapagliflozin and Metformin in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Alone
Brief Title: A Study of Prusogliptin Tablets Combined With Dapagliflozin Tablets and Metformin Hydrochloride Extended Release Tablets in Type 2 Diabetes
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HA1118-015
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Double-blind, Parallel-controlled
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Prusogliptin, Dapagliflozin(high dose), plus metformin XR (Experimental)
  Interventions: Drug: Prusogliptin, Dapagliflozin(high dose), Dapagliflozin (low dose) placebo, plus metformin XR
- Dapagliflozin(high dose), plus metformin XR (Active Comparator)
  Interventions: Drug: Prusogliptin placebo, Dapagliflozin(high dose), Dapagliflozin (low dose) placebo, plus metformin XR
- Prusogliptin, Dapagliflozin(low dose), plus metformin XR (Experimental)
  Interventions: Drug: Prusogliptin, Dapagliflozin(high dose) placebo, Dapagliflozin (low dose), plus metformin XR
- Dapagliflozin(low dose), plus metformin XR (Active Comparator)
  Interventions: Drug: Prusogliptin placebo, Dapagliflozin (high dose) placebo, Dapagliflozin (low dose), plus metformin XR
- Prusogliptin, plus metformin XR (Active Comparator)
  Interventions: Drug: Prusogliptin, Dapagliflozin (high dose) placebo, Dapagliflozin(low dose) placebo, plus metformin XR

INTERVENTIONS:
Drug: Prusogliptin, Dapagliflozin(high dose), Dapagliflozin (low dose) placebo, plus metformin XR — Prusogliptin, Dapagliflozin(high dose) and Dapagliflozin (low dose) placebo, once a day, 1 tablet per dose; Metformin XR, Once a day, the dosage remains the same as the pre-screening dose.
  Arms: Prusogliptin, Dapagliflozin(high dose), plus metformin XR
Drug: Prusogliptin placebo, Dapagliflozin(high dose), Dapagliflozin (low dose) placebo, plus metformin XR — Prusogliptin placebo, Dapagliflozin (high dose), Dapagliflozin (low dose) placebo, once a day, 1 tablet per dose; Metformin XR, Once a day, the dosage remains the same as the pre-screening dose
  Arms: Dapagliflozin(high dose), plus metformin XR
Drug: Prusogliptin, Dapagliflozin(high dose) placebo, Dapagliflozin (low dose), plus metformin XR — Prusogliptin, Dapagliflozin (high dose) placebo, Dapagliflozin (low dose), once a day, 1 tablet per dose; Metformin XR, Once a day, the dosage remains the same as the pre-screening dose
  Arms: Prusogliptin, Dapagliflozin(low dose), plus metformin XR
Drug: Prusogliptin placebo, Dapagliflozin (high dose) placebo, Dapagliflozin (low dose), plus metformin XR — Prusogliptin placebo, Dapagliflozin (high dose) placebo, Dapagliflozin (low dose), once a day, 1 tablet per dose; Metformin XR, Once a day, the dosage remains the same as the pre-screening dose
  Arms: Dapagliflozin(low dose), plus metformin XR
Drug: Prusogliptin, Dapagliflozin (high dose) placebo, Dapagliflozin(low dose) placebo, plus metformin XR — Prusogliptin, Dapagliflozin (high dose) placebo, Dapagliflozin (low dose) placebo, once a day, 1 tablet per dose; Metformin XR, Once a day, the dosage remains the same as the pre-screening dose
  Arms: Prusogliptin, plus metformin XR

SUMMARY:
This study is a multicenter, randomized, double-blind, parallel-controlled, phase III clinical trial to evaluate efficacy and safety of the triple combination therapy of prusogliptin, dapagliflozin and metformin in subjects with type 2 diabetes who have inadequate glycemic control on metformin alone.

DETAILED DESCRIPTION:
Avoid duplicating information that will be entered elsewhere, such as Eligibility Criteria or Outcome Measures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes was confirmed at least 10 weeks prior to the screening;
* Male or female, 18 years ≤ age ≤ 75 years;
* Body Mass Index (BMI) ≥ 18.5 kg/m^2, and ≤40 kg/m^2;
* Stable metformin therapy for at least 10 weeks prior to screening at a dose ≥ 1500 mg per day;
* The glycated hemoglobin must meet the following standards:During screening: 7.5% ≤ HbA1c ≤ 11.0% (local laboratory);Before random sampling: 7.0% ≤ HbA1c ≤ 10.5% (central laboratory);
* Be able to understand and follow the test procedures, voluntarily participate in the test and sign the ICF.

Exclusion Criteria:

* Type 1 diabetes or other special types of diabetes;
* ≥2 episodes of Grade 3 hypoglycemia within 6 months prior to screening, or any Grade 3 hypoglycemia occurring from screening to randomization;
* ≥1 episode of acute diabetic complications (e.g., diabetic ketoacidosis, hyperglycemic hyperosmolar state) within 6 months prior to screening or prior to randomization;
* Severe chronic diabetic complications (e.g., proliferative diabetic retinopathy, severe diabetic neuropathy, diabetic foot) within 6 months prior to screening;
* History of acute or chronic pancreatitis at screening or prior to randomization;
* Inflammatory bowel disease, partial intestinal obstruction, or chronic intestinal diseases associated with malabsorption within 6 months prior to screening or prior to randomization;
* Previous gastrointestinal surgeries that may cause malabsorption (excluding polypectomy and appendectomy), or chronic use of medications directly affecting gastrointestinal motility at screening or prior to randomization;
* Any cardiovascular event within 6 months prior to screening or prior to randomization, including: decompensated heart failure (NYHA Class III or IV); unstable angina, myocardial infarction, coronary artery bypass grafting, or coronary stent implantation; long QT syndrome or prolonged QTcF interval (male >450 ms, female >470 ms); clinically significant arrhythmia requiring treatment and deemed unsuitable for trial participation by the investigator;
* Hemorrhagic stroke or acute ischemic stroke within 6 months prior to screening or prior to randomization;
* Acute gallbladder disease within 6 months prior to screening, or active gallbladder disease requiring treatment at screening/prior to randomization;
* History of severe psychiatric disorders (e.g., depression, anxiety disorders), severe osteoporosis, or other medical conditions that may endanger participant safety as judged by the investigator;
* Malignancy (except clinically cured basal cell carcinoma or carcinoma in situ) diagnosed or treated within 5 years prior to screening or prior to randomization;
* Severe infection or trauma within 4 weeks prior to screening/prior to randomization; recurrent urinary tract infections or genital infections within 6 months prior to screening; or symptomatic urinary/genital infections at screening/prior to randomization;
* Clinically significant hematologic diseases (e.g., aplastic anemia, myelodysplastic syndrome) or conditions causing hemolysis or erythrocyte instability (e.g., malaria) at screening/prior to randomization;
* Pregnant or lactating women;
* Other conditions deemed unsuitable for trial participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 815 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-13 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in HbA1c at Week 24 | From baseline to week 24

SECONDARY OUTCOMES:
Proportion of participants with HbA1c of ≤6.5% and HbA1c of ≤7% at week 24 | From baseline to week 24
Relative change from baseline in HbA1c at week 12 | From baseline to week 12
Relative change from baseline in FPG at week 12 and week 24 | From baseline to week 12 and week 24
Relative change from baseline in 2h-PPG at week 12 and week 24 | From baseline to week 12 and week 24
Relative change from baseline in weight at week 12 and week 24 | From baseline to week 12 and week 24
Relative change from baseline in blood pressure at week 12 and week 24 | From baseline to week 12 and week 24
Relative change from baseline in blood lipid level at week 12 and week 24 | From baseline to week 12 and week 24
Relative change from baseline in 7-point blood glucose levels and average post-meal blood glucose increments at week 24 | From baseline to week 24
Proportion of participants who received rescue treatment after 24 weeks of treatment | From baseline to week 24

CONTACTS AND LOCATIONS:
Locations (1):
- No. 896, Zhongshan East Road, High-tech Industrial Development Zone, Shijiazhuang, Hebei, China